CLINICAL TRIAL: NCT07398443
Title: Using Novel Behavioral Economic Measures to Characterize Dual Marijuana and Tobacco Use in Young Adults
Acronym: MATEY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00000691; R01CA289409 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-06

CONDITIONS: Behavioral Economics; Cannabis Smoking; Tobacco Smoking
MeSH Terms: conditions — Marijuana Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cue Reactivity (Experimental): Participants will be exposed to neutral followed by cannabis or tobacco cues in a fixed sequence while they answer questions about their subjective state. The cues will include everyday items (e.g., eraser) and cannabis-related items (e.g., lighter).
  Interventions: Behavioral: Cue Reactivity

INTERVENTIONS:
Behavioral: Cue Reactivity — Participants will be exposed to neutral followed by cannabis or tobacco cues in a fixed sequence while they answer questions about their subjective state. The cues will include everyday items (e.g., eraser) and cannabis-related items (e.g., lighter).

SUMMARY:
The multi session experimental study aims to determine dual use patterns of marijuana and tobacco by assessing the impact of price and availability of marijuana and tobacco using a cross price elasticity of demand task. The study will recruit 120 non-treatment seeking emerging young adults (18-25 years) who smoke marijuana and tobacco.

DETAILED DESCRIPTION:
Young adulthood is a crucial time to study substance use disorders which increase cancer risk later in life. It is especially important to understand marijuana and tobacco use as most young adults often use both. Although dual use is related with increased long-term health and behavioral risks, underlying behavioral mechanisms remain unclear. This study aims to address this gap by using rigorous laboratory-based behavioral economic measure including a novel cross-price elasticity of demand (CPED) task and an innovative extension of cue-induced demand to assess cross-cue reactivity to better understand co- use. The results will help lead cessation efforts in this population and reduce cancer risk across the lifespan. Participants (N = 120) will be young adults (age 18-25) endorsing current tobacco and marijuana use and will complete 4 experimental in-person sessions. Following a phone-screen to assess preliminary eligibility, participants will come to the study center for in-person baseline screening. This screening consists of a urine toxicology screen, a breathalyzer test, and self-report questionnaires. The remaining three sessions will be completed in person which mainly consist of cross-cue reactivity sessions, self-report measures, and a qualitative exit interview following the final session.

ELIGIBILITY:
Inclusion Criteria:

1. Males/females who are 18 to 25 years of age
2. Young adults who currently smoke commercial tobacco cigarettes (≥1x weekly in the past 30 days and for the past six months)
3. Young adults who currently smoke marijuana (≥4 times in past 30 days and at least weekly on average for the last six months)
4. Participants must report purchasing their own tobacco and marijuana at least once in the past 6 months
5. Participants must speak, comprehend, and read English.

Exclusion Criteria:

1. Intention to quit marijuana or tobacco use in the next 30 days
2. Self-reported illicit drug or heavy episodic alcohol use on >20 days in the past month (excluding marijuana)
3. Individuals who are pregnant or breastfeeding
4. Positive saliva test for recent THC use
5. Breath alcohol level above 0 at any session.
6. Participants who exclusively roll their own tobacco cigarettes

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported cannabis craving | Up to 40 days post-baseline session
  This study utilizes a structured cannabis cue exposure paradigm. During cue exposure, participants rate subjective craving on a scale from 0, "Not at all," to 10, "Extremely." Cannabis craving will be assessed following neutral cue exposure and then cannabis cue exposure. The primary outcome will be change in cannabis craving.
Change in self-reported tobacco craving | Up to 40 days post-baseline session
  This study utilizes a structured tobacco cue exposure paradigm. During cue exposure, participants rate subjective craving on a scale from 0, "Not at all," to 10, "Extremely." Tobacco craving will be assessed following neutral cue exposure and then tobacco cue exposure. The primary outcome will be change in tobacco craving.

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No